CLINICAL TRIAL: NCT02732080
Title: Effect of Gradual Reperfusion on Myocardial Edema and Coronary Microvascular Integrity in Patients Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Gradual Versus Abrupt Reperfusion in Primary PCI (GUARD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Murat Sezer, Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 373
Record Dates: First submitted 2016-03-30; First posted 2016-04-08 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: ST-elevation Acute Myocardial Infarction
Keywords: primary percutaneous coronary intervention; microvascular obstruction; myocardial edema; microvascular resistance; acute myocardial infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deferred coronary stenting (Experimental): In this arm, after establishing TIMI -3 flow in infarct related artery with balloon angioplasty, patients will undergo stent implantation when coronary autoregulatory function was recovered (initial hyperemic flow was subsided and baseline resistance was increased). Recovery of the auto regulatory function will be determined by measuring microvascular flow and resistance. After stenting microvascular flow / resistance will continue to be monitored using pressure/flow sensor tipped guide wire until the completion of 1 hour follow up period.
  Interventions: Device: deferred coronary stenting
- Immediate stenting (Active Comparator): In this arm, patients will undergo stenting immediately after balloon angioplasty. After stent implantation, microvascular flow / resistance values will be continuously monitored using pressure/flow sensor tipped guide wire until the end of 1 hour follow up period.
  Interventions: Device: immediate stenting

INTERVENTIONS:
Device: deferred coronary stenting — Final coronary stenting will be performed when coronary auto regulation was recovered (approximately 30 minutes after establishment of TIMI III flow şn the infarct related artery)
  Arms: Deferred coronary stenting
Device: immediate stenting — Stent implantation will be performed immediately after balloon angioplasty (or thrombectomy or wire crossing) as it is performed in daily routine.
  Arms: Immediate stenting

SUMMARY:
After reopening of the infarct related artery by primary percutaneous coronary interventions (PPCI), microvascular damage at the related myocardial territory is not terminated immediately. This ongoing nature of microvascular damage leading to myocardial malperfusion is related to final infarct size. However, time course of the microvascular impairment /obstruction after PPCI in patients presented with ST-elevating acute myocardial infarction (STEMI) is not known. Routine primary percutaneous coronary interventions (PPCI) for ST-elevation acute myocardial infarction (STEMI) includes balloon angioplasty (or thrombectomy) followed immediately by stent implantation. However, stent implantation performed in this thrombotic setting may lead to a further microvascular damage by causing more distal embolisation and by inducing distal microvascular spasm by stretching the coronary vessel wall. Furthermore, sudden exposure of distal microcirculation to a high distal intracoronary pressure achieved by immediate stent implantation may exaggerate myocardial oedema which contributes microvascular damage substantially by external compression. However, results of studies investigating the efficacy of delayed stenting (24-48 hours later) in patients in whom TIMI -3 flow was achieved after balloon angioplasty were inconsistent.

In this study, STEMI patients undergoing PPCI, in whom epicardial reperfusion was achieved (TIMI-3 flow) by wire crossing or by balloon angioplasty or aspiration thrombectomy, will be randomised to immediate and delayed stenting groups. Delayed stenting will be performed at the time when coronary auto regulation was recovered which is going to be determined based on the continuous intracoronary hemodynamic monitoring after reperfusion.

DETAILED DESCRIPTION:
It was shown in ischemia/reperfusion models that after reopening of the occluded epicardial coronary artery, following initial hyperemic flow, myocardial blood flow in the area at risk rapidly and progressively declines and get stabilised approximately within 30 minutes.This finding implies that, in spite of the initial ischemic insult, coronary auto-regulation in the reperfused myocardial territory recovers. Nevertheless, this recovery requires some time after reperfusion was achieved. During total occlusion of an epicardial coronary artery, pre-arteriolar sphincters can be expected to be paralysed in widely open position in response to severely increased distal myocardial demand. Ischemic myocyte damage also contributes to malfunctioned pre-arteriolar sphincters. Therefore, full restoration of perfusion pressure distal to the infarct related artery by immediate stenting (direct or after angioplasty) may then fail to induce an immediate adaptive autoregulatory response (compensatory vasoconstriction) in the related microvascular territory, resulting in an inappropriately increased pressure in the damaged microcirculation. During total epicardial occlusion, ischemia/hypoxia induced damage and increased permeability at the capillary level lead to loss of structural integrity in the related microvascular territory. After immediate stenting, this severely damaged microcirculation is exposed to a suddenly increased uncontrolled intracoronary pressure which may consequently substantially contribute to intramyocardial haemorrhage and oedema.

Therefore, it was hypothesised that gradual reperfusion with delayed stenting performed when coronary auto regulatory function was recovered may lessen the myocardial oedema and/or haemorrhage by preventing/limiting uncontrolled increase in pressure in the distal microcirculation.

The recovery of coronary autoregulatory function in reperfused STEMI patients can be assessed by continuous monitoring of coronary (microvascular) blood flow and resistance values after restoration of epicardial blood flow by balloon angioplasty in individual basis.

In this study, following establishment of TIMI-3 flow by balloon angioplasty, patients will be randomized to immediate or delayed stenting groups. Continuous intracoronary hemodynamic monitorization will be performed in re-opened infarct related artery using a coronary guide wire equipped with pressure and flow sensors for a total of 1hour in both groups.

In delayed stent group, stent implantation will be performed in individual basis when coronary hemodynamic data indicates that coronary autoregulation was recovered (when initial hyperaemic flow response was subsided and baseline microvascular resistance was increased). Recovery of autoregulatory function will be determined by identification of stabilisation of baseline coronary flow velocity and baseline microvascular resistance in infarct related artery after balloon angioplasty. Stabilization will be decided by comparing basal coronary flow velocity and microvascular resistance values measured in non-infarct related coronary artery immediately before PPCI with the values that was being measured in re-opened infarct related artery. When baseline flow velocity and resistance values being recorded in IRA got close to the values measured in non-IRA, IRA will be stented. Intracoronary pressure and flow data will continuously be monitored until the end of 1 hour follow-up period.

In immediate stenting group, stent implantation will be performed immediately following angioplasty. Intracoronary pressure and flow data will continuously be monitored using dual sensor coronary guide wire until the end of 1 hour follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with ST-elevation acute myocardial infarction (STEMI) within 12 hours of their symptom onset in whom TIMI-3 flow was established in infarct related artery (IRA) after balloon angioplasty or thrombectomy.

Exclusion Criteria:

* Recanalized (TIMI I-III flow) IRA at coronary angiography.
* Patients in whom TIMI-3 flow was not able to be established after wire crossing, balloon angioplasty or thrombectomy.
* STEMI due to bypass-graft occlusion
* Severe heart failure or cardiogenic shock

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Coronary zero flow pressure (Pzf) | At the end of the 1 hour intracoronary hemodynamic monitorization

SECONDARY OUTCOMES:
Hyperemic microvascular resistance (HMR) | At the end of the completion of 1 hour intracoronary hemodynamic monitorization

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University, Istanbul Faculty of Medicine, Department of Cardiology, Istanbul
  - Istanbul University School of Medicine, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sezer M, Tas A, Demirtakan ZG, Broyd CJ, Ozcan A, Hasdemir H, Kocaaga M, Sezer I, Sonsoz MR, Atici A, Ozcan I, Umman B, Bugra Z, Davies JE, Escaned J, van Royen N, Umman S. Coronary microcirculation in nonculprit vessel territory in reperfused acute myocardial infarction. Microvasc Res. 2023 May;147:104495. doi: 10.1016/j.mvr.2023.104495. Epub 2023 Feb 3. PMID 36739961
- [Derived] Sezer M, Escaned J, Broyd CJ, Umman B, Bugra Z, Ozcan I, Sonsoz MR, Ozcan A, Atici A, Aslanger E, Sezer ZI, Davies JE, van Royen N, Umman S. Gradual Versus Abrupt Reperfusion During Primary Percutaneous Coronary Interventions in ST-Segment-Elevation Myocardial Infarction (GUARD). J Am Heart Assoc. 2022 May 17;11(10):e024172. doi: 10.1161/JAHA.121.024172. Epub 2022 May 16. PMID 35574948